CLINICAL TRIAL: NCT03767881
Title: A Multicenter, Prospective Study of EUS-Guided Transluminal Gallbladder Drainage in Patients With Acute Cholecystitis as an Alternative to Percutaneous Gallbladder Drainage
Brief Title: AXIOS™ for Gallbladder Drainage as an Alternative to Percutaneous Drainage IDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7108
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-11

CONDITIONS: Cholecystitis, Acute
Keywords: AXIOS; Acute Cholecystitis; Percutaneous Gallbladder Drainage; Cholecystitis; Gallbladder Drainage
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AXIOS(TM) Stent and Electrocautery Enhanced Delivery System (Experimental): Patients who are at high risk or unsuitable for surgery will receive an AXIOS stent under EUS guidance for treatment of acute cholecystitis.
  Interventions: Device: AXIOS(TM) Stent and Electrocautery Enhanced Delivery System

INTERVENTIONS:
Device: AXIOS(TM) Stent and Electrocautery Enhanced Delivery System — Patients who are at high risk or unsuitable for surgery will receive an AXIOS stent under EUS guidance for treatment of acute cholecystitis.

SUMMARY:
To evaluate the safety and effectiveness of the AXIOS™ Stent with Electrocautery Enhanced Delivery System in the management of symptoms of acute cholecystitis as an alternative to percutaneous gallbladder drainage.

DETAILED DESCRIPTION:
This study is a prospective, single arm, multi center trial. Treatment of up to 30 patients will take place at up to 9 clinical centers. Patients who meet all eligibility criteria will receive the AXIOS stent for up to 60 days indwell and 72 hour follow-up after stent removal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring intervention for the management of symptoms associated with acute cholecystitis
2. Patients referred for percutaneous drainage of the gallbladder who are not surgical candidates because of advanced age, anesthetic risk, significant co-morbidities and/or overall health
3. Eligible for endoscopic intervention
4. Acute Cholecystitis (AC) Grade I (mild) or II (moderate) per Tokyo guidelines:

   * AC Grade I (mild) defined as acute cholecystitis in an otherwise healthy patient with mild local inflammatory changes and without organ dysfunction. Criteria for grade II or III not met.
   * AC Grade II (moderate) defined by any one of the following characteristics

     * Leukocytosis (>18,000 cells per mm3)
     * Palpable, tender mass in right upper quadrant
     * Symptom duration >72 hours
     * Marked local inflammation (gangrenous or emphysematous cholecystitis, pericholecystic or hepatic abscess, biliary peritonitis)
5. Pre-drainage imaging confirms sufficient stone-free space to allow AXIOS™ stent deployment and complete flange expansion
6. 18 years of age or older
7. Willing and able to comply with the study procedures and patient or legally authorized representative (LAR) must provide written informed consent form (ICF) to participate in the study

Exclusion Criteria:

1. AC Grade III (severe) per Tokyo guidelines defined by organ dysfunction in any one of the following systems:

   * Cardiovascular - Hypotension requiring administration of ≥5μg/kg/min of dopamine or any dose of norepinephrine
   * Neurologic - decreased level of consciousness
   * Respiratory - PaO2/FiO2 <300
   * Renal - Oliguria and Creatinine >2.0 mg/dl (>177 μmol/liter)
   * Hepatic - International normalized ratio >1.5
   * Hematologic - Platelet count <100,000/mm3
2. Obvious signs on diagnostic imaging of perforated, extensive gangrenous or ischemic gallbladder
3. Hepatic abscess
4. Ascites
5. Patients with abnormal coagulation or who require ongoing complete anticoagulation
6. Bleeding diathesis
7. History of surgical treatment of acute cholecystitis (e.g. cholecystectomy)
8. Patients with a current percutaneous drainage
9. Patients with a history of percutaneous gallbladder drainage without AC free period following percutaneous drainage removal
10. Distance between gallbladder wall and duodenal or gastric wall > 1cm by US (ultrasound) at the time of drainage
11. Patients with intervening gastric varices or vessels within a one centimeter radius of the device insertion location
12. Patients that have allergies or are sensitive to any of the device materials
13. Patients with contraindications to use of electrical devices
14. Pregnancy
15. Prisoners and other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Irani, MBBS, MD, Principal Investigator — Virginia Mason Medical Center
Locations (7):
- United States (6):
  - University of Colorado Denver, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Parkview Medical Center, Fort Wayne, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Virginia Mason Medical Center, Seattle, Washington
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Irani SS, Sharma NR, Storm AC, Shah RJ, Chahal P, Willingham FF, Swanstrom L, Baron TH, Shlomovitz E, Kozarek RA, Peetermans JA, McMullen E, Ho E, van der Merwe SW. Endoscopic Ultrasound-guided Transluminal Gallbladder Drainage in Patients With Acute Cholecystitis: A Prospective Multicenter Trial. Ann Surg. 2023 Sep 1;278(3):e556-e562. doi: 10.1097/SLA.0000000000005784. Epub 2022 Dec 20. PMID 36537290

RESULTS

PARTICIPANT FLOW:
Groups:
- AXIOS Stent and Electrocautery Enhanced Delivery System: Patients will receive the AXIOS stent for the treatment of
  AXIOS: Patient will receive either transgastric or transduodenal endoscopic drainage for walled-off necrosis that are adherent to the gastric or bowel wall.
Period: Overall Study
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Started | 30
Completed | 25
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 10
  United States | 20
Weight [Mean (Standard Deviation); unit: kg] | 76.4 (17.8)
Height [Mean (Standard Deviation); unit: cm] | 168.6 (9.4)
BMI [Mean (Standard Deviation); unit: kg/m²] | 26.9 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Resolution of Acute Cholecystitis
Description: Time to resolution of acute cholecystitis measured in days. Resolution is defined as either a fever of less than 100.5°F, or at least a 4-point decrease in the pain score, or WBC count less than 12,000/cc, with improvement in at least two of these categories without the deterioration of the third category.
Time Frame: Up to 15 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AXIOS(TM) Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
days | 5.30 (14.90)
Statistical Analysis 1: Comparison: AXIOS(TM) Stent and Electrocautery Enhanced Delivery System; Test type: Non-Inferiority — The upper limit of a 97.8% confidence limit of the mean days to resolution of acute cholecystitis is compared to a Performance Goal of 3.5 days; t-test, 1 sided; Mean Difference (Final Values) = 3.5, 97.8% CI 1-sided [upper limit 10.78]

2. Secondary Outcome: Rate of Re-interventions
Description: Rate of re-interventions including but not limited to stent migration, stent occlusion by GB stones, and luminal debridement.
Time Frame: Through study completion, Up to 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
Participants | 5
Statistical Analysis 1: Comparison: AXIOS Stent and Electrocautery Enhanced Delivery System; Test type: Non-Inferiority — The upper limit of a 99.7% confidence limit of the proportion of patients with reintervention, including migration and occlusion, is compared to a Performance Goal of 46.2%; 1-sided Clopper-Pearson 99.7% CI; Performance Goal = 16.7, 99.7% CI 1-sided [upper limit 42.0]

3. Other Pre Specified Outcome: Stent Patency
Description: Stent patency (ability to facilitate gallbladder drainage) defined indirectly as resolution of acute cholecystitis or, in the absence of resolution of acute cholecystitis, endoscopic observation of unobstructed AXIOSTM stent lumen
Time Frame: Stent placement through stent removal, approximately 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 22
Participants | 22

4. Other Pre Specified Outcome: Number of Participants With Successful Technical Stent Placement.
Description: Technical AXIOS stent placement success, defined as transmural placement of the AXIOSTM stent with confirmed stent patency via (i) drainage visualized through the stent or fluoroscopically, or (ii) ability to endoscopically observe the inner walls of the gallbladder through the AXIOSTM stent
Time Frame: Intraoperative (stent placement)
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
Participants | 28

5. Other Pre Specified Outcome: Number of Participants With Successful Technical Stent Removal.
Description: Technical stent removal success, defined as the ability to remove the AXIOS stent endoscopically without stent removal related serious adverse events
Time Frame: Intraoperative (stent removal)
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 19
Participants | 19

6. Other Pre Specified Outcome: Acute Cholecystitis Recurrence
Description: Recurrence of acute cholecystitis and its management post AXIOS stent removal
Time Frame: Through study completion, up to 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
Participants | 3

7. Other Pre Specified Outcome: Number of Cumulative Hospital and ICU Days
Description: Number of cumulative hospital and ICU days from initial stent placement to resolution of symptoms of acute cholecystitis
Time Frame: Through study completion, up to 15 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 30
Days | 8.30 (7.14)

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
All-Cause Mortality (participants affected / at risk) | 5/30
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS Stent and Electrocautery Enhanced Delivery System (N=30)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Troponin T increased (Investigations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS Stent and Electrocautery Enhanced Delivery System (N=30)
Diarrhoea (Gastrointestinal disorders) | 9 (9)
C-reactive protein increased (Investigations) | 5 (6)
Urinary tract infection (Infections and infestations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03767881/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT03767881/SAP_001.pdf